CLINICAL TRIAL: NCT02278133
Title: A Phase Ib/II Multi-center, Open Label, Dose Escalation Study of WNT974, LGX818 and Cetuximab in Patients With BRAFV600-mutant KRAS Wild-type Metastatic Colorectal Cancer Harboring Wnt Pathway Mutations
Brief Title: Study of WNT974 in Combination With LGX818 and Cetuximab in Patients With BRAF-mutant Metastatic Colorectal Cancer (mCRC) and Wnt Pathway Mutations
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Array BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWNT974X2102C
Record Dates: First submitted 2014-10-06; First posted 2014-10-29 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic,; Colorectal cancer,; WNT974,; LGX818,; cetuximab,; BRAF-mutant,; mCRC,; BRAFV600-mutant,; KRAS
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — LGK974; encorafenib; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- WNT974, LGX818 and cetuximab combo (Experimental): Phase l: Dose Escalation phase; Phase ll: SIngle group assessing the triple combination of WNT974, LGX818 and cetuximab
  Interventions: Drug: WNT974; Drug: LGX818; Biological: Cetuximab

INTERVENTIONS:
Drug: WNT974
Drug: LGX818
Biological: Cetuximab

SUMMARY:
The purpose of this study is to assess the safety and anti-tumor activity of the triple combination of WNT974, LGX818 and cetuximab in BRAFV600-mutant mCRC with RNF43 mutations or RSPO fusions.

The design of this study is based upon the translational and pre-clinical data that suggest that Wnt pathway signals, increased due to RNF43 mutations or RSPO fusions, cooperate with the EGFR and BRAF signals to maintain the growth of BRAFV600 CRCs. Inhibition of these signals with the triple combination of WNT974, LGX818 and cetuximab may result in anti-tumor activity.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18 years
* Histological or cytological confirmed metastatic colorectal cancer
* Written documentation of KRAS wild-type status and BRAFV600-mutation with RNF43 mutation and/or RSPO fusion
* Progression of disease after at least one prior standard of care regimen or intolerant to irinotecan based regimens
* Availability of a representative tumor specimen (primary or metastatic, archival or newly obtained)
* Measurable disease as per RECIST v1.1
* Eastern cooperative oncology group (ECOG) performance status ≤ 2

Exclusion Criteria:

* Phase II only: Prior treatment with RAF inhibitors, Wnt pathway inhibitors, cetuximab, panitumumab, and/or other EGFR inhibitors
* Symptomatic brain metastasis. Patients previously treated or untreated for these conditions that are asymptomatic in the absence of corticosteroid and anti-epileptic therapy are allowed to enroll
* Current treatment with medications or consuming foods that are strong inhibitors or inducers of CYP3A4/5 or herbal medications and that cannot be discontinued at least one week prior to the start of treatment.
* Symptomatic or untreated leptomeningeal disease
* Acute or chronic pancreatitis
* Clinically significant cardiac disease
* Patients with any of the following laboratory values at Screening/baseline

  * Absolute neutrophil count (ANC) <1,500/mm3
  * Platelets < 100,000/mm3
  * Hemoglobin < 9.0 g/dL
  * Serum creatinine >1.5 x ULN or calculated or directly measured CrCl < 50% lower limit of normal
  * Serum total bilirubin >1.5 x ULN
  * AST/SGOT and/or ALT/SGPT > 2.5 x ULN, (> 5 x ULN if liver metastases present)
* Patients with impaired hepatic function as defined by Childs-Pugh class B or C
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral WNT974/LGX818

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-12; Primary Completion 2016-05-31 (Actual); Study Completion 2017-06-23 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities and exposure (AUC C1D15) to WNT974 and LGX818 (phase lb) | 12 months
  Phase Ib: To estimate the MTD(s) and/or RP2D(s) of the triple combination of WNT974, LGX818 and cetuximab in patients with BRAFV600-mutant, KRAS wild-type (WT) mCRC harboring upstream Wnt pathway mutations.
Overall response rate in phase II | 30 months
  Phase II: To estimate the preliminary anti-tumor activity of the RP2D(s) of the combination of WNT974, LGX818 and cetuximab in patients with BRAFV600-mutant metastatic CRC harboring upstream Wnt pathway mutations

SECONDARY OUTCOMES:
Overall response rate (ORR) (phase lb) | 36 months
  To assess additional parameters of clinical activity of WNT974 in combination with LGX818 and cetuximab in BRAFV600-mutant mCRC with evidence of upstream Wnt pathway activation.
Overall survival (OS) (phase lb/ll) | 36 months
  To assess additional parameters of clinical activity of WNT974 in combination with LGX818 and cetuximab in BRAFV600-mutant mCRC with evidence of upstream Wnt pathway activation.
Duration of response (DOR) (phase lb/ll) | 36 months
  To assess additional parameters of clinical activity of WNT974 in combination with LGX818 and cetuximab in BRAFV600-mutant mCRC with evidence of upstream Wnt pathway activation.
Time to response (TTR) (phase lb/ll) | 36 months
  To assess additional parameters of clinical activity of WNT974 in combination with LGX818 and cetuximab in BRAFV600-mutant mCRC with evidence of upstream Wnt pathway activation.
Progression free survival (PFS) (phase lb/ll) | 36 months
  To assess additional parameters of clinical activity of WNT974 in combination with LGX818 and cetuximab in BRAFV600-mutant mCRC with evidence of upstream Wnt pathway activation.
Disease control rate (DCR) (phase lb/ll) | 36 months
  To assess additional parameters of clinical activity of WNT974 in combination with LGX818 and cetuximab in BRAFV600-mutant mCRC with evidence of upstream Wnt pathway activation.
Plasma concentration of WNT974, LHA333, LGX818 (phase lb/ll) | 30 months
  To characterize the pharmacokinetics (PK) of WNT974, its pharmacologically active metabolite LHA333, and LGX818 when used in combination therapy with cetuximab
Number of participants with Adverse Events as a measure of safety and tolerability (phase lb/ll) | 30 months
  To characterize the safety and tolerability of WNT974 in combination with LGX818 and cetuximab in patients with BRAFV600-mutant mCRC with evidence of upstream Wnt pathway activation
Number of participants with Serious Adverse Events as a measure of safety and tolerability(phase lb/ll) | 30 months
  To characterize the safety and tolerability of WNT974 in combination with LGX818 and cetuximab in patients with BRAFV600-mutant mCRC with evidence of upstream Wnt pathway activation
Biomarker activations for WNT and RTK-MAPK pathways (phase Ib/II) | 32 months
  Phase Ib/II: To assess the pharmacodynamic effect of WNT974, LGX818 in combination with cetuximab and a potential relationship with clinical outcome
Number of participants with dose interruptions and dose reductions (phase Ib/II) | 30 months
  To characterize the safety and tolerability of WNT974 in combination with LGX818 and cetuximab in patients with BRAFV600-mutant mCRC with evidence of upstream Wnt pathway activation

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Call Center, Study Director — Array BioPharma, Inc.
Locations (18):
- United States (4):
  - Memorial Sloan-Kettering Cancer Center (MSKCC) MSKCC (3), New York, New York
  - Medical University of South Carolina Oncology Dept, Charleston, South Carolina
  - University of Texas/MD Anderson Cancer Center Onc. Dept,, Houston, Texas
  - University of Wisconsin / Paul P. Carbone Comp Cancer Center Univ Wisc, Madison, Wisconsin
- Array BioPharma Investigative Site, Parkville, Victoria, Australia
- Array BioPharma Investigative Site, Leuven, Belgium
- Canada (3):
  - Array BioPharma Investigative Site, Edmonton, Alberta
  - Array BioPharma Investigative Site, Vancouver, British Columbia
  - Array BioPharma Investigative Site, Toronto, Ontario
- France (2):
  - Array BioPharma Investigative Site, Bordeaux
  - Array BioPharma Investigative Site, Marseille
- Array BioPharma Investigative Site, Tel Aviv, Israel
- Array BioPharma Investigative Site, Milan, MI, Italy
- Array BioPharma Investigative Site, Amsterdam, Netherlands
- Array BioPharma Investigative Site, Singapore, Singapore
- Spain (3):
  - Array BioPharma Investigative Site, Barcelona, Catalonia
  - Array BioPharma Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Array BioPharma Investigative Site, Madrid

REFERENCES:
- [Derived] VAN Bussel MTJ, Bravenboer N, Essen HV, Snaebjornsson P, Appelman-Dijkstra NM, Schellens JH, Opdam FL. Bone Toxicity Case Report Combining Encorafenib, Cetuximab and WNT974 in a Phase I Trial. Anticancer Res. 2025 Jul;45(7):3137-3147. doi: 10.21873/anticanres.17677. PMID 40578933
- [Derived] Tabernero J, Van Cutsem E, Garralda E, Tai D, De Braud F, Geva R, van Bussel MTJ, Fiorella Dotti K, Elez E, de Miguel MJ, Litwiler K, Murphy D, Edwards M, Morris VK. A Phase Ib/II Study of WNT974 + Encorafenib + Cetuximab in Patients With BRAF V600E-Mutant KRAS Wild-Type Metastatic Colorectal Cancer. Oncologist. 2023 Mar 17;28(3):230-238. doi: 10.1093/oncolo/oyad007. PMID 36811382